CLINICAL TRIAL: NCT04625166
Title: Combi-elastography Assessment of Chronic Liver Disease Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Other Study IDs: S2020-387-01
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Non Alcoholic Fatty Liver; Hepatitis B; Drug-induced Liver Injury
Keywords: ultrasound; Elasticity Imaging Techniques
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hepatitis B; Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — liver tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
HITACH developed a new combi-elastography imaging technology combines shear wave imaging and strain imaging technology. In the study, not only the F index which is related to the stage of liver fibrosis can be obtained, but also the A index which is related to the stage of hepatitis can be obtained, which can not be obtained by other ultrasound devices.

DETAILED DESCRIPTION:
HITACHI developed a new combi-elastography imaging technology combines shear wave imaging and strain imaging technology to make full use of these two imaging modalities and make full use of different physical characteristics for imaging and quantitative analysis.

In the study, not only the F index which is related to the stage of liver fibrosis can be obtained, but also the A index which is related to the stage of hepatitis can be obtained, which can not be obtained by other ultrasound devices.

This technology is non-invasive, painless, simple and reliable, therefore it is bound to contribute to the early diagnosis of chronic liver disease and the real-time evaluation in the treatment process, which will play an important role in the clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis B:18-80 years old, no gender limit;Patient with chronic hepatitis B was diagnosed by liver histopathological examination;The pathological examination of liver tissue clearly provides G/S classification information. If there is steatosis, classification information is required;Patients without prehepatic ascites;Sign informed consent.
* Patients with MAFLD:18-80 years old, no gender limit;Meet the diagnostic criteria for metabolic-related fatty liver disease:Liver histological examination has liver steatosis,and meet one of the following three criteria,that is, overweight/obesity,type 2 diabetes (T2DM) or abnormal metabolism;Liver histopathological examination provides information on the classification of liver cell steatosis, fibrosis, and inflammation clearly;Patients without prehepatic ascites;Sign informed consent;
* Patients with DILI:18-80 years old, no gender limit;Patients with drug-induced liver injury was diagnosed by liver histological examination;The pathological examination of liver tissue provides G/S classification information clearly,If there is liver cell steatosis, classification information is required;Patients without prehepatic ascites;Sign informed consent;
* Healthy volunteers:Aged 18 to 60,Gender not limited,BMI<25;No abnormal signs by clinical examination,no fatty liver, No history of chronic liver disease such as hepatitis and liver cirrhosis, no serious gastrointestinal disease;Without metabolic syndrome;There is no history of long-term medication,do not taking any drugs before a month when checking;Did not find the primary lesions of liver, laboratory examination and clinical diagnosis without any liver disease and liver function is normal;Sign the informed consent.

Exclusion Criteria:

* Patients with chronic hepatitis B:Merging other disease caused by chronic liver disease (such as other types of viral hepatitis, drug-induced liver injury, autoimmune liver disease, alcoholic liver disease, metabolic related);Merging other systems' serious illness can't cooperate with elastic imaging checking (such as heart failure, renal failure,mental illness);Patients after liver transplantation;Pregnancy patients.
* Patients with MAFLD:Did/ongoing systemic chemotherapy patients;Patients with hepatic steatosis because of alcoholic liver disease,Viral hepatitis,Drug-induced liver disease,Autoimmune hepatitis or hepatolenticular degeneration et al;Special fatty liver disease cases because of drugs, total parenteral nutrition, inflammatory bowel disease, celiac disease, hypothyroidism,Cushing's syndrome,β lipoprotein lack hematic disease,Lipid atrophic diabetes or Mauriac syndrome et al;Merging other systems serious illness can't cooperate with elastic imaging checking(such as heart failure, renal failure,mental illness) ; Patients after liver transplantation;Patients with pregnancy.
* Patients with DILI:Other reasons or combined with other reasons caused liver damage (such as viral hepatitis, autoimmune liver disease, alcoholic liver disease, metabolic related fatty liver disease);The liver local infection and systemic infection;Merging other systems serious illness can't cooperate with elastic imaging checking(such as heart failure, renal failure,mental illness) ; Patients after liver transplantation;Patients with pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are eligible for the inclusion criteria as well as the exclusion criteria are enrolled in this study to obtain their clinical information.
Sampling Method: Non-Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
F index | 15 minutes
  To study the correlation between F index and the degree of fibrosis in patients of chronic liver disease.
A index | 15 minutes
  To study the correlation between A index and the degree of hepatitis in patients of chronic liver disease.
ATT index | 15 minutes
  To study the correlation between ATT index and the degree of steatosis in patients of metabolic associated fatty liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China